CLINICAL TRIAL: NCT02359058
Title: Phase 1b Study of Ramucirumab in Combination With Fluoropyrimidines and Platinum-Based Agents in Japanese Patients With Metastatic Gastric/Gastroesophageal Junction Adenocarcinoma
Brief Title: A Study of Ramucirumab Combination Therapy in Japanese Participants Who Have Advanced Stomach Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15532; I4T-JE-JVCX (Other: Eli Lilly)
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2017-07

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Ramucirumab; Capecitabine; Cisplatin; S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ramucirumab + Capecitabine + Cisplatin (Other): Ramucirumab (8 milligram per kilogram (mg/kg) given intravenously (IV) on days 1 and 8 in combination with 1000 mg/square meter (m^2) capecitabine given orally twice a day on days 1 through 14 and 80 mg/m^2 cisplatin given IV on day 1 of each 21 day cycle (up to 6 cycles). Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab; Drug: Capecitabine; Drug: Cisplatin
- Ramucirumab + S-1 + Cisplatin (Other): Ramucirumab 8 mg/kg given IV on days 1 and 8 of 21 day in combination with 40 mg/m^2 tegafur/gimeracil/oteracil (S-1) given orally twice a day on days 1 through 21 and 60 mg/m^2 cisplatin given IV on day 8 of each 35 day cycle (up to 8 cycles). Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab; Drug: Cisplatin; Drug: S-1
- Ramucirumab + S-1 + Oxaliplatin (Other): Ramucirumab 8 mg/kg given IV on days 1 and 8 in combination with 40 mg/m^2 S-1 given orally twice a day on days 1 through 14 and 100 mg/m^2 oxaliplatin given IV on day 1 of each 21 day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab; Drug: S-1; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806; IMC-1121B
Drug: Capecitabine — Administered orally
  Arms: Ramucirumab + Capecitabine + Cisplatin
Drug: Cisplatin — Administered IV
  Arms: Ramucirumab + Capecitabine + Cisplatin; Ramucirumab + S-1 + Cisplatin
Drug: S-1 — Administered orally
  Arms: Ramucirumab + S-1 + Cisplatin; Ramucirumab + S-1 + Oxaliplatin
Drug: Oxaliplatin — Administered IV
  Arms: Ramucirumab + S-1 + Oxaliplatin

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and antitumor response of ramucirumab in combination with platinum/fluoropyrimidine regimens in Japanese participants with advanced gastric/gastrooesophageal junction cancer who have not received chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* A histopathologically or cytologically confirmed diagnosis of gastric or gastroesophageal junction (GEJ) adenocarcinoma which is metastatic or locally advanced and unresectable. A participant with esophageal cancer is not eligible.
* Not have received prior first-line systemic chemotherapy for locally advanced and unresectable and/or metastatic disease. Participants whose disease has progressed after >6 months following the last dose of systemic treatment in the adjuvant/neoadjuvant setting are eligible.
* Measurable or nonmeasurable, but evaluable, disease, determined using guidelines in Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1 at the time of enrollment.
* The participant has adequate organ function.
* Resolution to Grade ≤1 by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; version [v]4.03) of all clinically significant toxic effects of prior locoregional therapy, surgery, or other anticancer.
* Female participants of childbearing potential must have a negative serum or urinary pregnancy. Have an estimated life expectancy of ≥12 weeks in the judgment of the investigator.

Exclusion Criteria:

* A significant bleeding disorder, vasculitis, or had a significant bleeding episode from the gastrointestinal tract within 12 weeks prior to enrollment.
* Uncontrolled arterial hypertension, despite standard medical management.
* A serious or nonhealing wound or peptic ulcer or bone fracture at enrollment.
* Undergone major surgery within 28 days prior to enrollment, or subcutaneous venous access device (reservoir) placement within 7 days prior to enrollment.
* Radiation therapy within 14 days prior to enrollment.
* Received any previous systemic therapy (including investigational agents) targeting vascular endothelial growth factor (VEGF) or the VEGF receptor signaling pathways.
* Cirrhosis at a level of Child-Pugh B (or worse); or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis.
* A serious illness or medical condition(s).
* Pregnant or breastfeeding.
* Dysphagia for oral medication.
* Known allergy or hypersensitivity to any study treatment.
* Human epidermal growth factor receptor (HER) 2 status of positive.
* Received treatment within 28 days of the initial dose of study drug with an investigational product or non-approved use of a drug or device.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- Japan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician, Osaka

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were considered completed if they either completed Cycle 1 of study drug or discontinued study drug due to a dose limiting toxicity (DLT) during Cycle 1.
Groups:
- Ramucirumab + Capecitabine + Cisplatin: Ramucirumab 8 mg/kg given intravenously (IV) on days 1 and 8 in combination with 1000 mg/square meter (m^2) capecitabine given orally twice a day on days 1 through 14 and 80 mg/m^2 cisplatin given IV on day 1 of each 21 day cycle (up to 6 cycles). Participants may continue to receive treatment until discontinuation criteria are met.
Period: Overall Study
Arm/Group | Ramucirumab + Capecitabine + Cisplatin | Ramucirumab + S-1 + Cisplatin | Ramucirumab + S-1 + Oxaliplatin
Started | 6 | 6 | 6
Received at Least 1 Dose of Study Drug | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramucirumab + Capecitabine + Cisplatin | Ramucirumab + S-1 + Cisplatin | Ramucirumab + S-1 + Oxaliplatin | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (10.93) | 60.3 (7.06) | 62.7 (6.98) | 60.2 (8.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 0 | 10
  Male | 2 | 0 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 6 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: Clinically significant events were defined as serious adverse events (SAE). A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: First Dose to Study Completion Plus 30-Day Safety Follow-Up (Up To 22 Months)
Population: All enrolled participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Capecitabine + Cisplatin | Ramucirumab + S-1 + Cisplatin | Ramucirumab + S-1 + Oxaliplatin
Number analyzed (Participants) | 6 | 6 | 6
Participants | 1 | 2 | 2

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) of Ramucirumab
Description: Maximum Serum Concentration (Cmax) of Ramucirumab.
Time Frame: Day 1, Day 8, Day 43, Day 50, Day 85 and Day 92: End of Infusion
Population: All enrolled participants who received at least one dose of the study drug and had evaluable ramucirumab PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | Ramucirumab + Capecitabine + Cisplatin | Ramucirumab + S-1 + Cisplatin | Ramucirumab + S-1 + Oxaliplatin
Number analyzed (Participants) | 6 | 6 | 6
microgram per milliliter (μg/mL)
  Day 1: number analyzed (Participants) | 6 | 5 | 6
  Day 1 | 149 (21) | 139 (23) | 137 (20)
  Day 8: number analyzed (Participants) | 6 | 6 | 5
  Day 8 | 229 (24) | 200 (21) | 211 (11)
  Day 43: number analyzed (Participants) | 4 | 3 | 3
  Day 43 | 205 (24) | 253 (11) | 180 (28)
  Day 50: number analyzed (Participants) | 3 | 5 | 3
  Day 50 | 273 (24) | 249 (24) | 207 (12)
  Day 85: number analyzed (Participants) | 2 | 3 | 1
  Day 85 | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of Cmax = 149.00 μg/mL, 216.00 μg/mL. | 272 (29) | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual value of Cmax = 239.00 μg/mL.
  Day 92: number analyzed (Participants) | 2 | 4 | 2
  Day 92 | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of Cmax = 191.00 μg/mL, 250.00 μg/mL. | 289 (22) | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of Cmax = 227.00 μg/mL, 278.00 μg/mL.

3. Secondary Outcome: Pharmacokinetics (PK): Minimum Serum Concentration (Cmin) of Ramucirumab
Description: Minimum Serum Concentration (Cmin) of Ramucirumab.
Time Frame: Day 8, Day 22, Day 29, Day 43, Day 50, Day 64, Day 71, Day 85, Day 92 and Day 106: Pre-Dose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable ramucirumab PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Ramucirumab + Capecitabine + Cisplatin | Ramucirumab + S-1 + Cisplatin | Ramucirumab + S-1 + Oxaliplatin
Number analyzed (Participants) | 6 | 6 | 6
μg/mL
  Day 8 | 43.8 (16) | 51.6 (28) | 43.2 (30)
  Day 22: number analyzed (Participants) | 4 | 6 | 5
  Day 22 | 40.9 (21) | 63.9 (33) | 41.8 (37)
  Day 29: number analyzed (Participants) | 5 | 5 | 5
  Day 29 | 84.6 (24) | 105 (19) | 81.6 (28)
  Day 43: number analyzed (Participants) | 5 | 4 | 5
  Day 43 | 60.8 (27) | 87.6 (34) | 68.5 (41)
  Day 50: number analyzed (Participants) | 4 | 5 | 3
  Day 50 | 91.7 (32) | 91.3 (28) | 86.2 (17)
  Day 64: number analyzed (Participants) | 3 | 4 | 3
  Day 64 | 47.7 (31) | 85.4 (34) | 81.5 (11)
  Day 71: number analyzed (Participants) | 4 | 4 | 3
  Day 71 | 71.1 (34) | 109 (13) | 124 (5)
  Day 85: number analyzed (Participants) | 4 | 4 | 2
  Day 85 | 55.5 (34) | 102 (18) | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of Cmin = 94.50 μg/mL, 98.00 μg/mL.
  Day 92: number analyzed (Participants) | 4 | 4 | 2
  Day 92 | 97.6 (24) | 119 (14) | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of Cmin = 66.00 μg/mL, 114.50 μg/mL.
  Day 106: number analyzed (Participants) | 3 | 3 | 2
  Day 106 | 68.6 (52) | 118 (12) | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of Cmin = 102.25 μg/mL, 107.50 μg/mL.

4. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response Rate)
Description: Objective response rate (ORR) was defined as the percentage of randomized participants achieving a best confirmed overall response of CR or PR using Response Evaluation Criteria in Solid Tumors (RECIST v1). CR was defined as the disappearance of all target and non-target lesions. PR was defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions, taking as reference the baseline sum LD and no progression in non-target lesions.
Time Frame: First Dose to Date of Objective Progressive Disease or Death Due to Any Cause (Up To 22 Months)
Population: All enrolled participants who received at least one dose of study drug and with measurable disease.
Measure: Number; unit: Percentage of participants
Groups:
- Total: Ramucirumab + Capecitabine + Cisplatin, Ramucirumab + S-1 + Cisplatin and Ramucirumab + S-1 + Oxaliplatin.
Arm/Group | Ramucirumab + Capecitabine + Cisplatin | Ramucirumab + S-1 + Cisplatin | Ramucirumab + S-1 + Oxaliplatin | Total
Number analyzed (Participants) | 5 | 1 | 5 | 11
Percentage of participants | 20 | 100 | 60 | 45.5

5. Secondary Outcome: Number of Participants With Treatment Emergent Anti-Ramucirumab Antibodies (TE-ADA)
Description: Number of participants with positive treatment emergent anti-ramucirumab antibodies was summarized by treatment group.
Time Frame: First dose to study completion plus 30-day safety follow-up (Up To 22 Months)
Population: All enrolled participants who received at least one dose of the study drug and had evaluable immunogenicity data.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Capecitabine + Cisplatin | Ramucirumab + S-1 + Cisplatin | Ramucirumab + S-1 + Oxaliplatin
Number analyzed (Participants) | 6 | 6 | 6
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose to study completion plus 30-day safety follow-up (Up To 22 Months)
Arm/Group | Ramucirumab + Capecitabine + Cisplatin | Ramucirumab + S-1 + Cisplatin | Ramucirumab + S-1 + Oxaliplatin
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 2/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Capecitabine + Cisplatin (N=6) | Ramucirumab + S-1 + Cisplatin (N=6) | Ramucirumab + S-1 + Oxaliplatin (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Capecitabine + Cisplatin (N=6) | Ramucirumab + S-1 + Cisplatin (N=6) | Ramucirumab + S-1 + Oxaliplatin (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 3 (3) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (8) | 1 (1) | 2 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (4)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 5 (12) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (5) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 5 (11) | 3 (4)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (4) | 2 (2)
Fatigue (General disorders) | 1 (1) | 3 (4) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (5)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (3) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Angular cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 5 (15) | 2 (5)
Platelet count decreased (Investigations) | 0 (0) | 3 (4) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 1 (2) | 2 (9) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (5) | 6 (17) | 3 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 3 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 4 (5) | 2 (3)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular pain (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.